CLINICAL TRIAL: NCT00452920
Title: A Phase I/II Study of Docetaxel as a Radiosensitizer for Locally Advanced Cervical Cancer (GIA 13026)
Brief Title: Docetaxel and Radiation Therapy in Treating Patients With Stage II, Stage III, or Stage IV Cervical Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 20020358; SCCC-2002058 (Other: University of Miami Institutional Review Board); WIRB-20050719 (Other: Western Insitutional Review Board)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Cervical Cancer
Keywords: cervical squamous cell carcinoma; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Docetaxel; Cesium-137; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Radiation: cesium Cs 137
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Docetaxel may make tumor cells more sensitive to radiation therapy. Giving docetaxel together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of docetaxel when given together with radiation therapy and to see how well they work in treating patients with stage II, stage III, or stage IV cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended phase II dose (RPTD) of docetaxel when administered with radiotherapy in patients with stage IIB-IVA cervical cancer. (Phase I)
* Assess the progression-free survival of patients treated with this regimen. (Phase II)

Secondary

* Determine the safety, feasibility, and toxicity of this regimen in these patients. (Phase I)
* Assess the toxicity of this regimen at the RPTD in these patients. (Phase II)
* Determine the response in patients treated with this regimen. (Phase II)

OUTLINE: This is a phase I, nonrandomized, prospective, dose-escalation study of docetaxel followed by an open-label phase II study.

* Phase I: Patients receive docetaxel IV over 30 minutes on day 1. Treatment repeats weekly for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo concurrent pelvic external-beam radiotherapy (EBRT) once daily 5 days a week for 5 weeks. Beginning 1-2 weeks after completion of EBRT, patients receive one or two applications of intracavitary low-dose-rate brachytherapy (LDR BT) comprising cesium-137.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose (RPTD) is the dose below the MTD.

* Phase II: Patients receive docetaxel at the RPTD, EBRT, and LDR BT as in phase I.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the uterine cervix

  * Locally advanced (stage IIB- IVA) disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* WBC ≥ 3,000/mm^3
* Creatinine normal
* Bilirubin normal
* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN) if alkaline phosphatase (AP) ≤ ULN OR AP ≤ 4 times ULN if SGOT and SGPT ≤ ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 6 months after completion of study treatment
* No history of severe allergic reactions to agents containing polysorbate 80
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude compliance with study requirements
* No peripheral neuropathy ≥ grade 2
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior unrelated therapy and recovered
* No prior chemotherapy or pelvic radiotherapy
* No other concurrent investigational agents or anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (Phase I)
Progression-free survival (Phase II)

SECONDARY OUTCOMES:
Response (Phase II)
Toxicity (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Lucci, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States